CLINICAL TRIAL: NCT02671890
Title: Expansion Cohort Study of Disulfiram and Chemotherapy in Pancreas Cancer Patients
Brief Title: Disulfiram and Chemotherapy in Treating Patients With Refractory Solid Tumors or Metastatic Pancreatic Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1512; R01CA195473 (NIH); NCI-2016-00007 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 15-003194 (Other: Mayo Clinic Institutional Review Board); MC1512 (Other: Mayo Clinic)
Record Dates: First submitted 2016-01-29; First posted 2016-02-02 (Estimated); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Pancreatic Adenocarcinoma; Refractory Malignant Solid Neoplasm; Stage IV Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Drug Therapy; Disulfiram; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort I (gemcitabine hydrochloride and disulfiram) (Experimental): Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15 and disulfiram PO on days 1-28 or days 1-35.
  Interventions: Drug: Disulfiram; Drug: Gemcitabine Hydrochloride; Other: Laboratory Biomarker Analysis
- Cohort II (chemotherapy and disulfiram) (Experimental): Patients receive chemotherapy at the discretion of the treating oncologist and disulfiram PO on days 1-28 or days 1-35.
  Interventions: Drug: Chemotherapy; Drug: Disulfiram; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Chemotherapy
  Other Names: Chemo; Chemotherapy (NOS); Chemotherapy, Cancer, General
  Arms: Cohort II (chemotherapy and disulfiram)
Drug: Disulfiram — Given PO
  Other Names: Antabuse; DS; Tetraethylthioperoxydicarbonic Diamide; Teturamin; TTD
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; FF 10832; FF-10832; FF10832; Gemcitabine HCI; Gemzar; LY-188011; LY188011
  Arms: Cohort I (gemcitabine hydrochloride and disulfiram)
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This partially randomized phase I trial studies the side effects and best dose of disulfiram when given together with chemotherapy in treating patients with a solid tumor that does not respond to treatment (refractory) or pancreatic cancer that has spread to other places in the body (metastatic) and to compare whether disulfiram and chemotherapy may reduce tumor induced muscle loss. Weight loss occurs in pancreatic cancer patients and is common in a multitude of other cancers. Patients with metastatic cancer and weight loss sometimes are not able to receive treatment due to physical weakness or debility. Disulfiram is a potential inhibitor of muscle degradation and may reduce tumor induced muscle wasting. Disulfiram may also help chemotherapy work better by making tumor cells more sensitive to the drug. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether giving chemotherapy with or without disulfiram is a better treatment for refractory solid tumors or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the maximally tolerated dose (MTD) of the combination of disulfiram and gemcitabine (gemcitabine hydrochloride) in unresectable solid tumor cancer patients (Cohort 1).

SECONDARY OBJECTIVES:

I. To describe the adverse event profile associated with this combination of disulfiram and chemotherapy (Cohort 2).

II. To describe changes in muscle area at the L3 level from baseline to 28 to 60 days from the baseline computed tomography (CT) scan in patients treated with disulfiram/chemotherapy and with placebo/chemotherapy (Cohort 2).

III. To describe changes in fist-grip strength from baseline to 28 to 35 days of treatment with disulfiram/gemcitabine and with placebo/chemotherapy (Cohort 2).

IV. To describe overall survival of pancreas cancer patients who disulfiram/chemotherapy or placebo/chemotherapy (Cohort 2).

V. To estimate the response rate per Response Evaluation Criteria in Solid Tumors (RECIST) criteria around 1 month post-treatment in patients who receive disulfiram/chemotherapy and placebo/chemotherapy (Cohort 2).

CORRELATIVE OBJECTIVE:

I. To assess the effect of disulfiram and chemotherapy on the ubiquitin proteasome and autophagy pathways within muscle, as assessed by means of muscle biopsies performed at baseline and after 28 to 35 days of treatment (Cohort 2) (this is for Mayo only patients and can be waived upon permission from the principal investigator [PI]).

OUTLINE: This is a phase I, dose-escalation study of disulfiram.

COHORT I: Patients receive gemcitabine hydrochloride intravenously (IV) over 30 minutes on days 1, 8, and 15 and disulfiram orally (PO) on days 1-28 or days 1-35.

COHORT II: Patients receive chemotherapy at the discretion of the treating oncologist and disulfiram PO on days 1-28 or days 1-35.

After completion of study treatment, patients are followed up at 30 days, and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1 (dose escalation): histologic or cytologic proof of any solid tumor that is incurable with no standard therapy that is likely to make a major impact on clinical outcomes
* Cohort 2 (MTD) only: metastatic adenocarcinoma of the pancreas; prior systemic treatment for metastatic disease is allowed
* Cohort 2 (MTD) only: Patient is thought to be a short- or long-term candidate for chemotherapy in the opinion of the treating oncologist
* Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 7 days prior to registration)
* Platelet >= 100,000/ mm^3 (obtained =< 7 days prior to registration)
* Total bilirubin =< 2 x upper limit of normal (ULN) (obtained =< 7 days prior to registration)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 3 x ULN (obtained =< 7 days prior to registration)
* Creatinine =< 1.5 x ULN (obtained =< 7 days prior to registration)
* Hemoglobin >= 9.0 g/dL (obtained =< 7 days prior to registration)
* Cohort 2 (MTD) only: prothrombin time (PT)/international normalized ratio (INR) =< 1.5 x ULN (only if muscle biopsy has not been waived, does not apply to non-Mayo sites that will not be conducting biopsies) (obtained =< 7 days prior to registration)
* Ability to provide written informed consent
* Life expectancy >= 12 weeks
* Cohort 2 (MTD) only: patient willing to undergo muscle biopsies at baseline and after 28 to 35 days of disulfiram/chemotherapy as required by the protocol unless the muscle biopsy has been waived after discussion with the principal investigator (PI); muscle biopsies will not be required at non-Mayo Clinic sites
* Cohort 2 (MTD) only: patient willing to have paraffin-embedded slides of the primary pancreas tumor or metastatic site, if available, sent to Mayo investigators for this study
* For women of childbearing potential only: negative urine or serum pregnancy test done =< 7 days prior to registration
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Able to swallow or have medication administered through a gastrostomy tube (G-tube) and absorb the medication
* Patient willing to complete a medication diary
* Patient agrees to use acceptable form of contraception during the study and for up to 30 days after last study drug dose if female partner is of childbearing potential

  * Acceptable forms of contraception:

    * Latex condom (always used with spermicide)
    * Diaphragm (always used with spermicide)
    * Cervical cap (always used with spermicide)
  * Acceptable forms of secondary contraception, when used along with a barrier method:

    * Hormonal contraception methods, including pills, patches, rings, or injections except progestin-only containing pills (i.e. "Mini-pill")
    * Tubal ligation
    * Partner's vasectomy
    * Intrauterine device (non-progesterone T)
    * Vaginal sponge (containing spermicide)
  * Other acceptable forms:

    * 100% commitment to abstinence
  * Unacceptable forms of contraception for women of childbearing potential:

    * Oral contraception containing progestins only
    * Intrauterine device (IUD) progesterone T
    * Female condom
    * Natural family planning (rhythm method) or breastfeeding
    * Fertility awareness
    * Withdrawal
    * Cervical shield

Exclusion Criteria:

* Known standard therapy for the patient's disease that is potentially curative
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, including localized infections, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric illness/social situations that would limit compliance with study requirements
* Untreated brain metastases
* Any of the following:

  * Pregnant women
  * Nursing women This study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown.
* Other concurrent chemotherapy, immunotherapy, radiotherapy, any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation) or receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Baseline of grade 2 or worse peripheral sensory neuropathy
* Receiving phenytoin
* Unable to abstain from alcohol for the duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-02-25 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) (Cohort I) | 28 days
  MTD is defined as the dose level below the lowest dose that induces dose limiting toxicity (DLT) in at least one-third of patients (at least 2 of a maximum of 6 new patients).

SECONDARY OUTCOMES:
Adverse events profile (Cohort I and II) | Up to 30 days post-treatment
  The number and severity of all adverse events (overall, by dose-level, and by tumor group) will be tabulated and summarized in this patient population. The grade 3+ adverse events will also be described and summarized in a similar fashion. This will provide an indication of the level of tolerance for this treatment combination in this patient group.
Toxicity profile defined as adverse events that are classified as either possibly, probably, or definitely related to study treatment (Cohorts I and II) | Up to 30 days post-treatment
  Non-hematologic toxicities will be evaluated via the ordinal Common Terminology Criteria (CTC) standard toxicity grading. Hematologic toxicity measures of thrombocytopenia, neutropenia, and leukopenia will be assessed using continuous variables as the outcome measures (primarily nadir) as well as categorization via CTC standard toxicity grading. Overall toxicity incidence as well as toxicity profiles by dose level, patient and tumor site will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses.
Overall survival (OS) (Cohort I and II) | From registration until death due to any cause, assessed up to 3 years
  OS will be summarized descriptively using the Kaplan-Meier estimate up to 3 years of follow-up in all alive patients.
Change in muscle area at the L3 level using a computed tomography (CT) scan (Cohort II) | Baseline to day 28
  Changes will be described using summary statistics and graphical techniques. A grayscale pixel histogram of the remaining muscle in the image will be constructed and summed. The number of pixels will then be converted to an area measurement in squared centimeters. All measurements and calculations for each image will be undertaken by two independent study personnel, and the average will be used in the analyses. A Wilcoxon rank sum test may be used as appropriate to compare percent changes of biomarkers between the muscle clinical responders and the non-responders based on CT scan measurements of muscle.
Response rate (Cohort II) | At 1 month post-treatment
  Response rate will be assessed using standard Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria.
Change in muscle area at the L3 level using a computed tomography scan (Cohort II) | Baseline to day 35
  Changes will be described using summary statistics and graphical techniques. A grayscale pixel histogram of the remaining muscle in the image will be constructed and summed. The number of pixels will then be converted to an area measurement in squared centimeters. All measurements and calculations for each image will be undertaken by two independent study personnel, and the average will be used in the analyses. A Wilcoxon rank sum test may be used as appropriate to compare percent changes of biomarkers between the muscle clinical responders and the non-responders based on CT scan measurements of muscle.
Changes in fist-grip strength as measured by hand dynamometer (Cohort II) | Baseline to day 28
  Changes will be described using summary statistics and graphical techniques. Patients will use 3 successive tries, and the average value will be used.
Changes in fist-grip strength as measured by hand dynamometer (Cohort II) | Baseline to day 35
  Changes will be described using summary statistics and graphical techniques. Patients will use 3 successive tries, and the average value will be used.

OTHER OUTCOMES:
Change in muscle protein expression level of total and phosphorylated (phosph)-signal transducer and activator of transcription 3 (STAT3) via immunohistochemistry | Baseline to up to 35 days
  Changes will be made at baseline and 28 to 35 days.
Changes in muscle messenger ribonucleic acid (mRNA) levels via real-time polymerase chain reaction | Baseline to up to 35 days
  Changes in mRNA transcripts of the muscle ubiquitin proteasome system (atrogin and muscle-specific RING finger protein 1) and STAT3 target genes (suppressor of cytokine signaling 3 and early growth response 1) will be made at baseline and 28 to 35 days.

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (2):
- United States (2):
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials